CLINICAL TRIAL: NCT03332940
Title: An Evaluation of the Safety of Intravenous (IV) Tc 99m Tilmanocept and a Comparison of Localization to Tc 99m Sulfur Colloid in Subjects With Nonalcoholic Steatohepatitis (NASH) and Healthy Controls (HC)
Brief Title: Safety Evaluation of IV Tc 99m Tilmanocept and Comparison of Imaging With Sulfur Colloid in Subjects With and Without NASH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No meaningful differences in the pattern of liver uptake were observed between Tc 99m tilmanocept and the comparator (Tc 99m sulfur colloid) after a review of the first six subjects.
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-30
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2023-01

CONDITIONS: Nonalcoholic Steatohepatitis; NASH - Nonalcoholic Steatohepatitis
Keywords: Tc99m-tilmanocept; Tilmanocept; NASH; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Technetium Tc 99m Sulfur Colloid; technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NASH subjects (Experimental): All subjects will receive a single IV injection of unfiltered sulfur colloid radiolabeled with 8 mCi Tc99m on study day 0. All subjects will receive a single IV injection of 200 mcg tilmanocept radiolabeled with 8 mCi Tc99m on study day 3.
  Interventions: Drug: Tc 99M Sulfur Colloid; Drug: Tc99m-tilmanocept
- Healthy controls (Experimental): All subjects will receive a single IV injection of unfiltered sulfur colloid radiolabeled with 8 mCi Tc99m on study day 0. All subjects will receive a single IV injection of 200 mcg tilmanocept radiolabeled with 8 mCi Tc99m on study day 3.
  Interventions: Drug: Tc 99M Sulfur Colloid; Drug: Tc99m-tilmanocept

INTERVENTIONS:
Drug: Tc 99M Sulfur Colloid — Sulfur colloid is a radiotracer that is indicated for imaging areas of functional reticuloendothelial cells in the liver, spleen, and bone marrow.
  Other Names: Sulfur colloid
Drug: Tc99m-tilmanocept — Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Other Names: Tilmanocept; Lymphoseek

SUMMARY:
This is a prospective, open-label, multicenter, safety, comparative study of IV administered Tc99m-tilmanocept and unfiltered Tc99m sulfur colloid in the detection of and assessment of three dimensional tessellation localization to the liver in subjects with and without moderate to severe nonalcoholic steatohepatitis (NASH) by planar and SPECT/CT imaging.

This study is designed to evaluate the safety and tolerability of Tc99m-tilmanocept in subjects with NASH.

ELIGIBILITY:
Inclusion Criteria:

* ALL SUBJECTS:

  1. The subject has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) authorization before the initiation of any study-related procedures.
  2. The subject is ≥18 years of age at the time of consent.
  3. The subject has a body mass index (BMI) between 18 and 45.

     CONTROL SUBJECTS:
  4. The subject is deemed to be clinically free of any infectious/inflammatory disease(s) for at least 4 weeks prior to the consent date.
  5. The subject has not taken any antibiotics for at least 4 weeks prior to the consent date.

NASH SUBJECTS:

4. The subject has biopsy-confirmed NASH within 12 months prior to enrollment. 5. The subject has a NAFLD Activity Score (NAS) of ≥ 4, with a score of at least 1 for each steatosis, lobular inflammation, and hepatocyte ballooning.

6. The subject has fibrosis staging of F3-F4.

Exclusion Criteria:

* ALL SUBJECTS:

  1. The subject is pregnant or lactating.
  2. The subject size or weight is not compatible with imaging per the investigator.
  3. The subject has received radiation therapy or chemotherapy or has a previous diagnosis of cancer other than basal cell carcinoma.
  4. The subject has renal insufficiency as demonstrated by a GFR of < 60 mL/min.
  5. The subject has a chronic or persistent infection or has any condition that would, in the opinion of the examining physician, preclude their participation.
  6. The subject has a known allergy to or has had an adverse reaction to dextran exposure.
  7. The subject has received an investigational product within 30 days prior to the Tc 99m sulfur colloid administration.
  8. The subject has received any radiopharmaceutical within 7 days prior to the administration of Tc 99m sulfur colloid.
  9. The subject is HIV positive.
  10. The subject has a history of alcohol abuse or currently consumes alcohol in excess of 3 drinks/day for men or 2 drinks/day for women.
  11. The subject has hepatitis B or C.

      CONTROL SUBJECTS:
  12. The subject has hepatic insufficiency as demonstrated by ALT (alanine aminotransferase [SGPT]) or AST (aspartate aminotransferase [SGOT]) greater than two times the upper limit of normal (ULN).
  13. The subject has been diagnosed with NASH, NAFLD, or other chronic liver disease.
  14. The subject has been diagnosed with metabolic syndrome or Type I or II diabetes.

NASH SUBJECTS:

12. The subject has any chronic liver disease aside from NASH/NAFLD.

13. The subject has uncontrolled diabetes as indicated by an A1c >9% within the 3 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Adverse Drug Reaction | 5 days after Tc 99m tilmanocept injection
  Proportion of subjects experiencing noxious pharmacologic activity/an Adverse Drug Reaction (ADR).

SECONDARY OUTCOMES:
Localization of Tc 99m tilmanocept | 5 days after Tc 99m tilmanocept injection
  Determine the three dimensional tessellation localization of Tc 99m tilmanocept by planar and SPECT/CT imaging in subjects with NASH and asymptomatic controls.
Localization of Tc 99m sulfur colloid | 5 days after Tc 99m tilmanocept injection
  Determine the three dimensional tessellation localization of unfiltered Tc 99m sulfur colloid by planar and SPECT/CT imaging in subjects with NASH and asymptomatic controls.
Localization Distribution Comparison | 5 days after Tc 99m tilmanocept injection
  Comparison of liver localization distribution tessellation pattern intensities between Tc 99m tilmanocept and unfiltered Tc 99m sulfur colloid.

OTHER OUTCOMES:
Tc 99m tilmanocept Localization Distribution of SPECT/CT vs Elastography | 5 days after Tc 99m tilmanocept injection
  Concordance of intrahepatic localization tessellation discrimination of Tc 99m tilmanocept (intrahepatic disease heterogeneity) by SPECT/CT imaging and elastography.
Tc 99m sulfur colloid Localization Distribution of SPECT/CT vs Elastography | 5 days after Tc 99m tilmanocept injection
  Concordance of intrahepatic localization tessellation discrimination of Tc 99m sulfur colloid (intrahepatic disease heterogeneity) by SPECT/CT imaging and elastography.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Navidea Biopharmaceuticals, Inc.
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cope FO, Abbruzzese B, Sanders J, Metz W, Sturms K, Ralph D, Blue M, Zhang J, Bracci P, Bshara W, Behr S, Maurer T, Williams K, Walker J, Beverly A, Blay B, Damughatla A, Larsen M, Mountain C, Neylon E, Parcel K, Raghuraman K, Ricks K, Rose L, Sivakumar A, Streck N, Wang B, Wasco C, Williams A, Schlesinger LS, Azad A, Rajaram MVS, Jarjour W, Young N, Rosol T, McGrath M. Corrigendum to the inextricable axis of targeted diagnostic imaging and therapy: An immunological natural history approach [Nucl Med Biol 43 (2016) 215-225]. Nucl Med Biol. 2016 Dec;43(12):837. doi: 10.1016/j.nucmedbio.2016.10.001. No abstract available. PMID 27866590
- [Background] Cope, F.O., W. Metz, et al. Innovations in receptor-targeted precision imaging at Navidea: diagnosis up close and personal. Nature Outlook (31 October 2013); S125-S129.
- See also: Navidea Biopharmaceuticals, Inc. — https://www.navidea.com/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT03332940/Prot_SAP_000.pdf